CLINICAL TRIAL: NCT00470171
Title: Efficacy and Safety of Ursodesoxycholic Acid in the Management of Non-Alcoholic Steatohepatitis
Brief Title: Pilot Study of Ursodesoxycholic Acid in Non-Alcoholic Steatohepatitis
Acronym: URSONASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axcan Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URSONASH05-01; EudraCT n° : 2005-001931-31
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Serum Levels of ALAT Transaminases; Serum Markers for Fibrosis and Hepatic Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ursodesoxycholic acid

SUMMARY:
This is a phase II study with direct individual benefit. It is a randomized, double blind placebo controlled study whose aim is to evaluate the efficacy and tolerance of ursodesoxycholic acid in patients who have been diagnosed with non-alcoholic steatohepatitis.

The hepatoprotective effects of ursodesoxycholic acid may ameliorate the hepatic impairment associated with non-alcoholic steatohepatitis leading to subsequent significant decreases in transaminase elevations and non-invasive markers for hepatic fibrosis A positive response is defined as a significantly larger decrease in average ALAT levels between the time of inclusion in the study and the end of the treatment for the ursodesoxycholic acid group as compared to the placebo group.

The duration of the study will be 12 months. An end of treatment evaluation (EoT) will take place at the end of the 12th month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* Hepatic biopsy consistent with non-alcoholic steatohepatitis: presence of >20% steatosis associated with hepatocyte swelling and/or intralobular necrosis within the last 18 months.
* Serum levels of ALAT and/or ASAT > 50 UI/L at the time of screening (with at least 3 elevated transaminase values within the last 12 months).

Exclusion Criteria:

* Hepatic biopsy not performed within the last 18 months.
* A single normal transaminase value within the last 12 months.
* Treatment with ursodesoxycholic acid within the last 12 months.
* Loss of more than 15% body weight between the time of the liver biopsy and the time of screening.
* Alcohol consumption of >20 g/day for women and > 30 g/day for men
* Hepatitis from other causes: chronic viral hepatitis B or C, elevated ferritin levels associated with C282Y homozygosity, primary biliary cirrhosis, primary sclerosing cholangitis, well documented auto-immune hepatitis (specific autoantibodies, hypergammaglobulinemia, consistent histologic changes), alpha1 antitrypsin deficiency, Wilson's disease, HIV infection.
* NASH from secondary causes: long term amiodarone administration, corticosteroid therapy, anti-obesity surgery within the last 2 years, tamoxifen.
* Child's type B or C cirrhosis.
* Presence of hepatocellular carcinoma.
* Treatment with rosiglitazone or pioglitazone currently or during the 3 preceding years, treatment with Vitamin E within the 6 months prior to screening.
* Women who are pregnant or nursing.
* Unavailability of hepatic biopsy slides for centralized interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
A positive response is defined as a significantly larger decrease in average ALAT levels between the time of inclusion in the study and the end of the treatment for the ursodesoxycholic acid group as compared to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Ratziu, M.D., Ph.D., Principal Investigator — La Pitié Salpétrière Hospital, Paris, France
Locations (1):
- La Pitié Salpétrière Hospital, Paris, France